CLINICAL TRIAL: NCT03211364
Title: Comparing Mobilization Techniques for the Hemiplegic Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/0404
Record Dates: First submitted 2017-06-13; First posted 2017-07-07 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Hemiplegic Shoulder; Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients do not know what are the intervention techniques or what is the control technique.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Angular mobilization (Active Comparator): Angular mobilization of the shoulder joint in the frontal plane.
  Interventions: Other: Glenohumeral mobilization
- Angular mobilization with soft tissue techniques (Active Comparator): Angular mobilization performed in the scapular plane. Additional soft tissue techniques to eliminate limitations created by tensed muscles in order to perform capsular stretch.
  Interventions: Other: Glenohumeral mobilization
- Scapular mobilization (Placebo Comparator): Scapular mobilization without glenohumeral movement.
  Interventions: Other: Scapular mobilization

INTERVENTIONS:
Other: Glenohumeral mobilization — Comparing the effect of angular mobilization in frontal or scapular plane and of providing soft tissue techniques on hemiplegic shoulder range of motion and pain.
  Arms: Angular mobilization; Angular mobilization with soft tissue techniques
Other: Scapular mobilization
  Arms: Scapular mobilization

SUMMARY:
One of the main complications after stroke is hemiplegic shoulder pain. It is known that one of the most frequent causes of hemiplegic shoulder pain is a restricted range of motion in the shoulder joint. Therefore, it is necessary to preserve the passive range of motion by using the most optimal mobilization technique. The aim of this study is to compare 2 different techniques in order to document their influence on shoulder range of motion and shoulder pain in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Upper limb impairment

Exclusion Criteria:

* Shoulder pain on the hemiplegic side with onset before the stroke
* Surgery at the hemiplegic shoulder
* Active movement possible within the whole range of motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Range of motion of the shoulder using goniometry | Measuring every 4 weeks up to 12 weeks after admission to the study protocol
  Range of motion of the shoulder joint is measured using a goniometer
Shoulder pain using visual analogue scale | Measuring every 4 weeks up to 12 weeks after admission to the study protocol
  Shoulder pain during rest, night and activities by using visual analogue scale (0-10)

SECONDARY OUTCOMES:
Spasticity of the shoulder muscles using the Modified Ashworth Scale | Measuring every 4 weeks up to 12 weeks after admission to the study protocol
  Spasticity of upper limb muscles related to the shoulder using Modified Ashworth Scale
Trunk Impairment Scale to assess trunk stability | Measuring every 4 weeks up to 12 weeks after admission to the study protocol
  Trunk stability using the Trunk Impairment Scale
Fugl-Meyer Assessment - upper limb part to assess voluntary muscle activity | Measuring every 4 weeks up to 12 weeks after admission to the study protocol
  voluntary muscle activity upper limb using the upper limb part of the Fugl-Meyer Scale

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Cambier, Prof, Study Chair — University Ghent; Kristine Oostra, Dr, Principal Investigator — University Hospital, Ghent
Locations (1):
- Vakgroep Revaki - Ghent University, Ghent, Belgium